CLINICAL TRIAL: NCT02436681
Title: A Prospective Post-Market Clinical Evaluation of Miromatrix Biological Mesh for Hiatal Hernia Repair
Brief Title: Miromatrix Biological Mesh for Hiatal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miromatrix Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015002
Record Dates: First submitted 2015-05-04; First posted 2015-05-07 (Estimated); Results first posted 2019-09-18 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Hiatal Hernia
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MIROMESH (Other): Single-arm study. MIROMESH will be used in the surgical repair of hiatal hernias.
  Interventions: Device: MIROMESH

INTERVENTIONS:
Device: MIROMESH

SUMMARY:
Miromatrix Medical has developed MIROMESH® - a new, noncrosslinked, acellular mesh derived from the highly vascularized porcine liver. MIROMESH received FDA 510(k) clearance with an indication for reinforcement of soft tissue on March 31, 2014 under K134033. This study will serve to provide clinicians with high-quality clinical data in order to provide them with a higher degree of confidence when selecting MIROMESH for hiatal hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 80 years old on the day of study enrollment
* able and willing to sign the consent form and comply with all study visits and procedures
* able to undergo elective laparoscopic hiatal hernia repair
* free of cognitive or speech impairment
* documented, symptomatic type II or III hernia ≥5cm in the axial/vertical dimension
* commit to non-smoking for at least 4 weeks prior to procedure

Exclusion Criteria:

* previous operation of the esophagus or stomach
* sensitivity to porcine material
* pregnant or plan to be pregnant within next 2 years
* immunocompromised or at risk of immunosuppression (i.e. be HIV positive, be experiencing organ rejection, be a recent or anticipated chemotherapy recipient) as determined by the Investigator
* require emergent operation for acute gastric volvulus or strangulation
* American Society of Anesthesiology (ASA) class 4 or greater
* BMI ≥40
* life expectancy of less than 2 years at the time of enrollment
* associated gastrointestinal disease that requires extensive medical or surgical intervention that might interfere with the quality of life assessment (e.g. Crohn's disease)
* any condition in the opinion of the Investigator that would preclude the use of the study device, or preclude the subject from completing the follow-up requirements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rosen, M.D., Principal Investigator — The Cleveland Clinic
Locations (6):
- United States (6):
  - University of Kentucky, Lexington, Kentucky
  - Monmouth Medical Center, Long Branch, New Jersey
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Virginia Heartburn and Hernia Institute, Lorton, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from treating surgeon's normal practice.
Pre-assignment Details: 3 found to be ineligible (inclusion/exclusion) at surgery 2 Withdrew consent prior to surgery 2 Mesh not implanted per surgeon discretion 2 Canceled procedure
Groups:
- MIROMESH: MIROMESH was used for laparoscopic paraesophageal hernia repair
Period: Overall Study
Arm/Group | MIROMESH
Started | 41
Completed | 27
Not Completed | 14
Not completed — Lost to Follow-up | 10
Not completed — Withdrawal by Subject | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | MIROMESH
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 41
ASA Status [Count of Participants; unit: Participants]
  1 - Healthy Patients | 1
  2 - Mild to moderate systemic disease, controlled | 23
  3 - Severe disease process, limited activity | 14
  Unknown | 3
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.7 (4.0)
Smoking Status [Count of Participants; unit: Participants]
  Current | 1
  Ex-smoker | 11
  Never | 29
Gastroesophageal Reflux Disease Health Related Quality of Life (GERD-HRQL) [Mean (Standard Deviation); unit: Score] — The Gastroesophageal Reflux Disease Health Related Quality of Life (GERD-HRQL) scale assess on symptoms associated with gastroesophageal reflux disease. There are 10 questions (each representing a GERD symptom such as heartburn) answered on a 6-point scale of 0 - 6 with 0 indicating no symptoms and 5 indicating incapacitating symptoms. The answer to all questions are summed to give you a final score on the scale. Scores may range for 0 (no symptoms) to 50 (incapacitating symptoms).
  Score | 19.3 (13.5)
GERD-HRQL Global Assessment [Count of Participants; unit: Participants] — Global rating of how satisfied patients are with their condition.
  Participants
    Satisfied | 7
    Neutral | 3
    Dissatisfied | 29
    Unknown | 2
SF36 - Physical Component Summary Score [Mean (Standard Deviation); unit: Score] — The Short-Form 36 (SF-36) is a general health assessment tool comprised of 8 sub-scales including Physical Function, Role Physical, Bodily Pain, and General health which assess aspects of physical health. These are used to make an overall physical health score, the Physical Component Summary score (PCS). The higher the score the better the subject's physical health. Range from 0-100.
  Score | 41.5 (9.9)
SF36 - Mental Component Summary Score [Mean (Standard Deviation); unit: Score] — The Short-Form 36 (SF-36) is a general health assessment tool comprised of 8 sub-scales including Vitality, Role Emotional, Social Functioning, and Mental health which assess aspects of Mental health. These are used to make an overall mental health score, the Mental Component Summary score (MCS). The higher the score the better the subject's mental health. Range from 0-100.
  Score | 46.6 (12.0)
SF36 - Physical Functioning [Mean (Standard Deviation); unit: Score] — The Short-Form 36 (SF-36) is a general health assessment tool comprised of 8 sub-scales including Physical Functioning which assess aspects of physical health. The higher the score the better the subject's physical health. Range from 0-100.
  Score | 38.9 (9.5)
SF36 - Social Functioning [Mean (Standard Deviation); unit: Score] — The Short-Form 36 (SF-36) is a general health assessment tool comprised of 8 sub-scales including Social Functioning which assess aspects of mental health. The higher the score the better the subject's physical health. Range from 0-100.
  Score | 42.5 (10.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a Hernia Recurrence Requiring Reoperation
Description: Failure of the index hernia operation which requires another operative procedure to correct. Hernia recurrence was assessed with a barium upper gastrointestinal series or in some cases other imaging analysis to characterize the anatomy of the esophagus.
Time Frame: 2 years
Population: Lost to follow up 10 Withdrew Consent 2 Death 2
Measure: Count of Participants; unit: Participants
Arm/Group | MIROMESH
Number analyzed (Participants) | 27
Participants | 0

2. Other Pre Specified Outcome: Radiographic Recurrence
Description: Reports the number of radiographic recurrence of hernia that does not require surgery and are generally asymptomatic. Hernia recurrence was assessed with a barium upper gastrointestinal series or in some cases other imaging analysis to characterize the anatomy of the esophagus.
Time Frame: 2 years
Population: Lost to follow up 10 Withdrew Consent 2 Death 2
Measure: Count of Participants; unit: Participants
Arm/Group | MIROMESH
Number analyzed (Participants) | 27
Participants | 3

3. Other Pre Specified Outcome: GERD-HRQL
Description: The Gastroesophageal Reflux Disease Health Related Quality of Life (GERD-HRQL) scale assess on symptoms associated with gastroesophageal reflux disease. There are 10 questions (each representing a GERD symptom such as heartburn) answered on a 6-point scale of 0 - 6 with 0 indicating no symptoms and 5 indicating incapacitating symptoms. The answer to all questions are summed to give you a final score on the scale. Scores may range for 0 (no symptoms) to 50 (incapacitating symptoms).
Time Frame: 2 years
Population: Lost to follow up 10 Withdrew Consent 2 Death 2
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | MIROMESH
Number analyzed (Participants) | 27
Score | 3.8 (5.3)
Statistical Analysis 1: Comparison: MIROMESH; Test type: Superiority; p < 0.0001, t-test, 1 sided

4. Other Pre Specified Outcome: GERD-HRQL Global Assessment
Description: Same as baseline
Time Frame: 2 years
Population: Lost to follow up 10 Withdrew Consent 2 Death 2
Measure: Count of Participants; unit: Participants
Arm/Group | MIROMESH
Number analyzed (Participants) | 27
Participants
  Satisfied | 23
  Neutral | 2
  Dissatisfied | 1
  Unknown | 1

5. Other Pre Specified Outcome: SF36 - Physical Component Summary Score
Description: Measure Description: The Short-Form 36 (SF-36) is a general health assessment tool comprised of 8 sub-scales including Physical Function, Role Physical, Bodily Pain, and General health which assess aspects of physical health. These are used to make an overall physical health score, the Physical Component Summary score (PCS). The higher the score the better the subject's physical health. Range from 0-100.
Time Frame: 2 years
Population: Lost to follow up 10 Withdrew Consent 2 Death 2
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | MIROMESH
Number analyzed (Participants) | 27
Score | 47.2 (9.3)
Statistical Analysis 1: Comparison: MIROMESH; Test type: Superiority; p = 0.0468, t-test, 1 sided

6. Other Pre Specified Outcome: SF36 - Mental Component Summary Score
Description: Measure Description: The Short-Form 36 (SF-36) is a general health assessment tool comprised of 8 sub-scales including Vitality, Role Emotional, Social Functioning, and Mental health which assess aspects of Mental health. These are used to make an overall mental health score, the Mental Component Summary score (MCS). The higher the score the better the subject's mental health. Range from 0-100.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | MIROMESH
Number analyzed (Participants) | 27
Score | 53.6 (8.0)

7. Other Pre Specified Outcome: SF36 - Physical Functioning
Description: Measure Description: The Short-Form 36 (SF-36) is a general health assessment tool comprised of 8 sub-scales including Physical Functioning which assess aspects of physical health. The higher the score the better the subject's physical health. Range from 0-100.
Time Frame: 2 years
Population: Same as baseline
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | MIROMESH
Number analyzed (Participants) | 27
Score | 45.6 (10.6)
Statistical Analysis 1: Comparison: MIROMESH; Test type: Superiority; p = 0.014, t-test, 1 sided

8. Other Pre Specified Outcome: SF36 - Social Functioning
Description: Measure Description: The Short-Form 36 (SF-36) is a general health assessment tool comprised of 8 sub-scales including Social Functioning which assess aspects of mental health. The higher the score the better the subject's physical health. Range from 0-100.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | MIROMESH
Number analyzed (Participants) | 27
Score | 49.5 (8.8)
Statistical Analysis 1: Comparison: MIROMESH; Test type: Superiority; p = 0.018, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 2 years post procedure
Arm/Group | MIROMESH
All-Cause Mortality (participants affected / at risk) | 2/41
Serious Adverse Events (participants affected / at risk) | 2/41
Other Adverse Events (participants affected / at risk) | 10/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MIROMESH (N=41)
Acute respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Nausea/vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MIROMESH (N=41)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Edema at GE Junction (Gastrointestinal disorders) | 2 (2)
Food Bolus Obstruction (Gastrointestinal disorders) | 1 (1)
Acute Gastric Distension (Gastrointestinal disorders) | 1 (1)
Anterior Gastropexy Pain (Gastrointestinal disorders) | 1 (1)
Mild Hypoxia (Blood and lymphatic system disorders) | 1 (1)
Nausea and Vomiting (Gastrointestinal disorders) | 2 (2)
Pleural Effusion requiring drainage (General disorders) | 1 (1)
Soreness (General disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was not a randomized controlled trial, thus direct comparisons to no treatment or other treatment cannot be made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-05): https://cdn.clinicaltrials.gov/large-docs/81/NCT02436681/Prot_SAP_000.pdf